CLINICAL TRIAL: NCT06506500
Title: Unilateral Biportal Endoscopy Lumbar Interbody Fusion (ULIF) Versus Posterior Lumbar Interbody Fusion (PLIF) in Management of Single Level Lumbar Degenerative Disease: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-365-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Degenerative Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ULIF: Unilateral Biportal Endoscopy Lumbar Interbody Fusion
- PLIF: Posterior Lumbar Interbody Fusion

SUMMARY:
The study aimed to compare the clinical efficacy and safety of unilateral biportal endoscopic lumbar interbody fusion (ULIF) with posterior lumbar interbody fusion (PLIF) in the treatment of single-level lumbar degenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with lumbar disc herniation, lumbar spinal stenosis, or lumbar spondylolisthesis based on their medical history, physical signs, and imaging exams such as lumbar anteroposterior and lateral radiographs (including hyperextension and hyperflexion positions), lumbar CT, and lumbar MR. (2) The patient has clear indications for surgical treatment: ① Conservative treatment for more than three months has been ineffective or the symptoms have continued to worsen ② The patient's symptoms are severe and interfere with their daily work and life ③ The patient exhibits signs of cauda equina nerve compression (such as numbness in the perineal area, loss of bowel and bladder control, etc.).

(3) The patient is undergoing their initial single-segment ULIF or PLIF surgery at our hospital.

Exclusion Criteria:

1. Patients with lumbar degenerative diseases involving two or more segments
2. Pathological changes caused by other diseases, such as spinal infections, spinal trauma, spinal tumors, neurological diseases, etc.
3. Patients with lumbar spondylolisthesis exceeding Meyerding Grade II or degenerative scoliosis with a Cobb angle greater than 20 degrees
4. History of previous lumbar surgery
5. History of previous tumor disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients who have been diagnosed with lumbar disc herniation, lumbar spinal stenosis, or lumbar spondylolisthesis.
  2. The patient has clear indications for surgical treatment.
  3. The patient is undergoing their initial single-segment ULIF or PLIF surgery at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
ODI | before surgery，1-week，1-month，3-month，6-month and 1-year postoperative
  Oswestry Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University,, Guangzhou, Guangdong, China